CLINICAL TRIAL: NCT00744081
Title: Open-label Multicenter Trial of Glivec® (Imatinib Mesylate, Formerly Known as STI571) in Combination With Chemotherapy (MTC) in Patients With Refractory or Relapsed Acute Myeloid Leukemia (AML)
Brief Title: Imatinib + MTC in Relapsed / Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Lothar Bergmann, Principal Investigator, Goethe University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG-R1
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: AML
MeSH Terms: interventions — Imatinib Mesylate; Mitoxantrone; Topotecan

INTERVENTIONS:
Drug: Glivec
Drug: Mitoxantrone
Drug: Topotecan
Drug: AraC

SUMMARY:
The purpose of this study is to show superiority in complete responses of combination therapy MTC plus Glivec in patients with refractory or relapsed AML compared to a historical control which was treated with MTC alone.

ELIGIBILITY:
Inclusion Criteria:

* Refractory AML after primary therapy
* First relapse after a safe previous diagnosis of de novo or secondary AML
* Age > 18 years
* Serum bilirubin < 2.0 mg/dl
* Serum creatinine < 1.5 times the normal value or a creatinine clearance > 60 ml/min
* ECG and heart echography prior to start of therapy without severe findings
* Overall condition < 2 according to ECOG criteria
* Life expectancy > 6 weeks
* Written informed consent by patients with full legal capacity

Exclusion Criteria:

* Serious secondary disease (clinically relevant cardiac disease, chronic- obstructive pulmonary disease, hepatic dysfunction, renal insufficiency)
* Active secondary neoplasia (exception: adequately treated basalioma or epidermoid cancer and cervical carcinoma)
* Known hypersensitivity to topoisomerase-I inhibitors
* Overall condition > 2 according to ECOG criteria
* Pregnant/breast feeding women
* Serious intercurrent infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To show superiority in complete responses of combination therapy MTC plus Glivec in patients with refractory or relapsed AML compared to a historical control which was treated with MTC alone.

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Bergmann, MD, PhD, Study Chair — University Hospital of Frankfurt, Medical Dept. II
Locations (1):
- University of Frankfurt, Medical Dept. II, Frankfurt, Germany

REFERENCES:
- See also: (German Leukemia Trial Registry) — http://www.studienregister-online.de